CLINICAL TRIAL: NCT03084302
Title: Sedentary Behavior in Pregnancy and Cardiovascular Health: the Monitoring Movement and Health (MoM Health) Study
Brief Title: Monitoring Movement and Health Study
Acronym: MoM Health
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Bethany Barone Gibbs, PhD, University of Pittsburgh
Other Study IDs: PRO16120430
Record Dates: First submitted 2017-03-07; First posted 2017-03-20 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy Related; Obesity; Hypertension
Keywords: sedentary behavior; physical activity
MeSH Terms: conditions — Obesity; Hypertension; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Women in their first trimester of pregnancy, aged 18-45, who plan to receive their prenatal care from University of Pittsburgh Medical Center providers.

SUMMARY:
The investigators will study sedentary behavior (SED) across pregnancy in young women. We hypothesize that SED will increase across pregnancy and that higher SED will be related to worse cardiovascular health, specifically elevated blood pressure (BP) and excessive gestational weight gain (GWG). Pregnancy is a biologically relevant period during which CVD risk factors may develop or worsen, contributing to future CVD. Pregnant women also spend most of their day sedentary, which is defined as too much sitting as distinct from too little exercise. SED has emerged as a risk factor, independent from moderate-to-vigorous physical activity (e.g., exercise), for elevated BP, obesity, diabetes, CVD, and mortality in general populations, but there are no recommendations for SED during pregnancy and few studies evaluate SED across pregnancy. These few studies are limited by small sample size, lack of repeated measures across trimesters, suboptimal SED assessment methodology, and a failure to link with clinical outcomes (e.g., BP, GWG). The investigators will address these gaps in a prospective study that will measure SED in 130 pregnant women across three trimesters using state-of-the-art objective activity monitors capable of measuring min-by-min activity by both intensity and posture. We will also measure BP and GWG during each trimester and, further, will link to and abstract all prenatal clinic weights and BPs, glucose screening results, gestational diabetes, preeclampsia, and adverse birth outcomes. Lastly, with the long-term goal of identifying women at high risk of SED during pregnancy and designing effective interventions, the investigators will efficiently evaluate correlates and determinants of SED which have never been studied during pregnancy.

DETAILED DESCRIPTION:
Objective: The investigators aim to conduct a prospective cohort study using state-of-the-art, noninvasive measurement of sedentary behavior in n=130 pregnant women during each trimester of their first pregnancy. We will link sedentary behavior to gestational weight gain, blood pressure, and potential determinants such as demographics, health conditions and behaviors, psychosocial factors, perceptions/beliefs, and the environment.

Specific Aims:

Aim 1: Objectively measure sedentary behavior across pregnancy trimesters Aim 2: Relate objectively-measured sedentary behavior to blood pressure and gestational weight gain across pregnancy Aim 3: Characterize correlates and determinants of sedentary behavior during pregnancy

1.3 Background: Cardiovacular disease (CVD) remains the leading cause of death in women with minimal declines over the past 30 years among women <55 years old. Stagnant rates of CVD mortality in younger women have occurred alongside notable declines in men and older adults and are thought to be due, in part, to high rates of obesity and elevated blood pressure (BP). Related to this, the American Heart Association (AHA) recently identified primordial prevention, a population-level approach that targets preventing rather than treating CVD risk factors, as a necessary strategy to reduce the CVD burden. To achieve primordial prevention, the target must be populations at risk for developing CVD risk factors (vs. those with existing risk factors), such as younger women.

Pregnancy is a biologically unique period for young women during which CVD risk factors such as obesity and high blood pressure (BP) can develop or worsen, contributing to future CVD. Pregnant women also spend most of their time in sedentary behavior (SED). SED is any behavior that occurs in a seated/reclining position with low energy expenditure and is now recognized as a behavior that is distinct from inactivity, or a lack of moderate-vigorous physical activity (MVPA). Though MVPA has known benefits, SED is an emerging, independent risk factor for obesity, CVD, and mortality. Importantly, prolonged bouts of SED (accumulated in bouts lasting 30 min or more) in non-pregnant persons are more strongly related to obesity and induce unfavorable hemodynamic responses, such as increased BP. We hypothesize that too much SED across pregnancy is an important contributor to excess gestational weight gain (GWG) and elevated BP, two important CVD risk factors in young women.

Remarkably, a dearth of studies evaluates SED across pregnancy. In cross-sectional studies, pregnant women spend 50-60% of their day in SED and SED is highest in the 3rd trimester. Yet, no study has evaluated if SED increases across pregnancy (repeated measurements) using best practice SED assessment methodology (objective device capable of capturing posture and intensity). Moreover, no study has evaluated whether greater SED is associated with increased GWG and BP in pregnant women, which in turn are known to impact pregnancy health and later maternal CVD risk. Current guidelines only advise MVPA for pregnant women with no recommendations about SED, highlighting the research gaps about SED and its consequences during pregnancy. Moreover, clarifying the role of SED in pregnancy is important because lowering SED might be a feasible strategy for pregnant women, who have low participation in9 and unique barriers to MVPA. Lastly, little is known about correlates and determinants of SED in pregnancy. Such data are critical for identifying women at risk for high SED during pregnancy and for developing effective interventions.

1.4 Significance: Sedentary behavior is a novel risk factor for weight gain, high BP, and CVD, yet patterns, correlates, determinants and consequences of sedentary behavior are poorly understood in pregnant women. Sedentary behavior is the most common behavior in pregnant women, but the dearth of research studies applying state-of-the-art sedentary behavior assessment methods and with repeated measures across pregnancy is a major research gap that we intend to address with this proposal. To the investigators' knowledge, no studies with optimal sedentary behavior measurement, assessing both posture and intensity while awake (i.e., activPAL), have been conducted in pregnant women. Beyond this, few studies have evaluated temporal trends in sedentary time across gestation. There is no research examining bouts of extended, uninterrupted sedentary time which have particularly deleterious effects on BP and are more strongly related to high BMI. Lastly, correlates and determinants of sedentary behavior are poorly understood overall and, in particular, among pregnant women. Before effective interventions can be designed to reduce sedentary behavior in pregnancy, nonmodifiable and modifiable factors associated with sedentary behavior must be better understood. Thus, the objective, longitudinal measurement of sedentary behavior in pregnancy proposed in this application will determine patterns, correlates, determinants, and consequences of sedentary behavior in pregnancy to move toward future goals of 1) clarifying risks and whether sedentary behavior recommendations are appropriate for pregnant women, 2) identifying groups at risk for high sedentary behavior, and 3) informing intervention targets. Further, this research addresses the AHA's mission to reduce the burden of CVD by investigating a novel strategy for primordial prevention of cardiovascular disease in young women.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 weeks pregnant
* 18-45 years old
* plan to receive prenatal care and deliver with University of Pittsburgh Medical Center providers

Exclusion Criteria:

* use of medication to treat diabetes or hypertension
* medical condition that severely limits physical activity (e.g., cannot walk 2 blocks)
* other serious medical condition that could affect outcomes (such as systemic lupus, chronic renal disease, or hepatitis)

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: We will recruit 120 women in their first trimester of pregnancy. Women must be 18-45 and must be seeing a UPMC provider for their prenatal care and delivery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Barone Gibbs, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with secondary investigators after the following process. 1) Secondary investigators will submit a proposal to the principal investigator that will be reviewed by all Coinvestigators. 2) If all investigators approve, the secondary investigator will obtain institutional review board approval to conduct the proposed analyses, and 3) a deidentified dataset including only requested variables will be provided to the secondary researcher.
Time Frame: Data requests will be accepted 6 months after the study funding expired (September 2020).
Access Criteria: Outside investigators wishing to gain access to MoM Health data will be required to submit a document outlining the rationale and hypotheses to be tested, specific data requested, and analytic plan. This will be reviewed by MoM Health Study investigators for rigor and overlap of existing analyses. All reasonable requests will be honored.

REFERENCES:
- [Background] Barone Gibbs B, Paley JL, Jones MA, Whitaker KM, Connolly CP, Catov JM. Validity of self-reported and objectively measured sedentary behavior in pregnancy. BMC Pregnancy Childbirth. 2020 Feb 11;20(1):99. doi: 10.1186/s12884-020-2771-z. PMID 32046663
- [Result] Barone Gibbs B, Jones MA, Jakicic JM, Jeyabalan A, Whitaker KM, Catov JM. Objectively Measured Sedentary Behavior and Physical Activity Across 3 Trimesters of Pregnancy: The Monitoring Movement and Health Study. J Phys Act Health. 2021 Mar 1;18(3):254-261. doi: 10.1123/jpah.2020-0398. Epub 2021 Jan 28. PMID 33508775
- [Result] Jones MA, Catov JM, Jeyabalan A, Whitaker KM, Barone Gibbs B. Sedentary behaviour and physical activity across pregnancy and birth outcomes. Paediatr Perinat Epidemiol. 2021 May;35(3):341-349. doi: 10.1111/ppe.12731. Epub 2020 Oct 30. PMID 33124060
- [Result] Jones MA, Whitaker K, Wallace M, Barone Gibbs B. Demographic, Socioeconomic, and Health-Related Predictors of Objectively Measured Sedentary Time and Physical Activity During Pregnancy. J Phys Act Health. 2021 Jun 17;18(8):957-964. doi: 10.1123/jpah.2021-0097. Print 2021 Aug 1. PMID 34140419
- [Result] Whitaker KM, Zhang D, Kline CE, Catov J, Barone Gibbs B. Associations of Sleep With Sedentary Behavior and Physical Activity Patterns Across Pregnancy Trimesters. Womens Health Issues. 2021 Jul-Aug;31(4):366-375. doi: 10.1016/j.whi.2021.02.003. Epub 2021 Mar 11. PMID 33715925
- [Derived] Paley JL, Jones MA, Catov JM, Whitaker KM, Kozai AC, Barone Gibbs B. Associations of Physical Activity and Sedentary Behaviors with Depressive Symptoms and Mood Disturbance Throughout Pregnancy. J Womens Health (Larchmt). 2024 Aug;33(8):1128-1138. doi: 10.1089/jwh.2023.0419. Epub 2024 Feb 6. PMID 38324012
- [Derived] Gibbs BB, Jones MA, Whitaker KM, Ross ST, Davis KK. Measurement of Barriers, Attitudes, and Expectations for Sitting Less in Pregnancy. Am J Health Behav. 2021 Nov 15;45(6):956-970. doi: 10.5993/AJHB.45.6.1. PMID 34969408

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnant Women
Started | 120
Completed | 105
Not Completed | 15
Not completed — Miscarriage, twin pregnancy, congenital abnormality | 9
Not completed — No valid objective monitor data | 6

BASELINE CHARACTERISTICS:
Population: Participants with at least one valid trimester of activity data and without a miscarriage, congenital abnormality, or twin pregnancy.
Arm/Group | Pregnant Women
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 105
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 80
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Having High Sedentary Behavior (by Trajectory)
Description: Trajectories identified from objective data across trimesters. High sedentary behavior was defined as the highest group (~10.9 hr/day) based on growth mixture models from the objective data.
Time Frame: 1st, 2nd, and 3rd trimester of pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- Full Cohort: All participants with at least one valid objective data measure
Arm/Group | Full Cohort
Number analyzed (Participants) | 105
Participants | 45

2. Primary Outcome: Number of Participants Classified as Having Low Moderate-to-vigorous Intensity Physical Activity (by Trajectory)
Description: Low levels of physical activity across trimesters, identified by growth mixture modelling. The low trajectory corresponded to about 114 minutes per week or about 16 minutes per day.
Time Frame: 1st, 2nd, and 3rd trimester of pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- Full Cohort: All women with at least one valid assessment of objective activity or sedentary behavior data.
Arm/Group | Full Cohort
Number analyzed (Participants) | 105
Participants | 29

3. Secondary Outcome: Number of Participants With Excessive Gestational Weight Gain
Description: from study visits and medical records excessive gestational weight gain was defined using 2009 Institute of Medicine Guidelines (reference: Institute of Medicine and National Research Council. Weight gain during pregnancy: reexamining the guidelines. Washington, DC: The National Academies Press; 2009)
Time Frame: at delivery
Population: Women with at least one valid trimester of objective data and available medical records.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 100
Participants | 49

4. Secondary Outcome: Adverse Pregnancy Outcomes
Description: from study visits and medical records includes hypertensive disorders of pregnancy, preterm birth, intrauterine growth restrictions, gestational diabetes
Time Frame: during pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 100
Participants | 19

ADVERSE EVENTS:
Time Frame: During study participation (6 months)
Description: This study is observational. Only adverse events related to the minimal risk study procedures were collected.
Arm/Group | Full Cohort
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03084302/Prot_SAP_000.pdf